CLINICAL TRIAL: NCT00003730
Title: A Multicenter Randomized Trial, With Direct Individual Benefit, to Determine the Optimal Circadian Time of Vinorelbine Administration Combined With Chronomodulated Infusion of 5-Fluorouracil in Previously Treated Patients With Metastatic Breast Cancer
Brief Title: Vinorelbine Plus Fluorouracil in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-05971; EORTC-05971
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Vinorelbine

INTERVENTIONS:
Drug: fluorouracil
Drug: vinorelbine tartrate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized clinical trial to study the effectiveness of vinorelbine plus fluorouracil in treating women who have metastatic breast cancer that has been previously treated with at least one regimen of chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the least toxic time of vinorelbine administration when combined with chronomodulated fluorouracil in women with previously treated metastatic breast cancer.
* Determine the toxic effects and dose intensities of each drug in these women.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior chemotherapy (second line vs third line) and participating center. Patients are randomized to 1 of 8 vinorelbine dosing times (0000, 0300, 0600, 0900, 1200, 1500, 1800, or 2100).

Patients receive vinorelbine IV over 20 minutes on days 1 and 6 and fluorouracil IV over 12 hours according to a chronomodulated delivery rate (2200 to 1000 with a maximum dose at 0400) on days 1-4. Treatment repeats every 3 weeks for at least 3 courses in the absence of unacceptable toxicity.

Patients are followed for 30 days.

PROJECTED ACCRUAL: A minimum of 80 patients (10 per dosing time) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic breast cancer
* At least 1 line of prior chemotherapy for metastatic disease (adjuvant or neoadjuvant chemotherapy is considered first line if completed less than one year prior to palliative chemotherapy)
* No cerebral metastases
* Hormonal receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* Not specified

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm ^3

Hepatic:

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 1.58 mg/dL

Cardiovascular:

* No clinically significant cardiac insufficiency or ischemic disease

Pulmonary:

* No bronchoconstriction other than pulmonary lymphangitis

Other:

* No serious chronic disease
* No bowel obstruction
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy
* No concurrent prophylactic growth factor

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* No prior high-dose chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent hormonal therapy
* No concurrent steroid therapy except in an emergency

Radiotherapy:

* At least 4 weeks since prior radiotherapy (for primary tumor or axillary or mammary chain treatment only)
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No other concurrent antitumor therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 1998-12; Primary Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Coudert, MD, Study Chair — Centre Georges Francois Leclerc
Locations (17):
- Belgium (3):
  - VZW Monica Campus Eeuwfeestkliniek, Antwerp
  - C.H.C - Asbl, Liège
  - CHU Liege - Domaine Universitaire du Sart Tilman, Liège
- France (8):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Lutte Contre le Cancer Georges-Francois Leclerc, Dijon
  - Hopital Perpetuel Secours, Levallois-Perret
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Hopital Saint-Louis, Paris
  - Centre Rene Huguenin, Saint-Cloud
  - Hopital Bellevue, Saint-Etienne
  - Hopital Paul Brousse, Villejuif
- University Hospital of Heraklion, Iraklion (Heraklion), Crete, Greece
- Italy (5):
  - Istituto per la Ricerca e Cura del Cancro, Candiolo (Turin)
  - Ospedale San Carlo Borromeo, Milano (Milan)
  - Azienda Ospedale S. Luigi - Universita Di Turin, Orbassano, (Torino)
  - Fondazione Salvatore Maugeri, Pavia
  - Istituti Fisioterapici Ospitalieri - Roma, Rome

REFERENCES:
- [Result] Coudert B, Focan C, Genet D, Giacchetti S, Cvickovic F, Zambelli A, Fillet G, Chollet P, Amoroso D, Van Der Auwera J, Lentz MA, Marreaud S, Baron B, Gorlia T, Biville F, Levi F. A randomized multicenter study of optimal circadian time of vinorelbine combined with chronomodulated 5-fluorouracil in pretreated metastatic breast cancer patients: EORTC trial 05971. Chronobiol Int. 2008 Sep;25(5):680-96. doi: 10.1080/07420520802384036. PMID 18780198